CLINICAL TRIAL: NCT00003134
Title: A Phase II Trial of Irinotecan in Recurrent Glioma
Brief Title: Irinotecan in Treating Patients With Recurrent Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-967251; NCI-2012-02257 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000065900 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult oligodendroglioma; adult mixed glioma; adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Glioma; Astrocytoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: irinotecan (Experimental): Patients receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22. This is followed by a 2 week rest and continues for a maximum of 6 courses. Patients who received prior nitrosoureas, also receive reduced starting doses of irinotecan. The dosages may be increased once per patient after the first course if toxic effects are acceptable.
  Patients are followed every 3 months for the first year, every 6 months for the next 4 years, then annually until death.
  Interventions: Drug: irinotecan hydrochloride
- Arm II: irinotecan (Experimental): Patients receive irinotecan on day 1 every 3 weeks for up to 12 courses. Patients who received prior nitrosoureas receive reduced starting doses of irinotecan. The dosages may be increased once per patient after the first course if toxic effects are acceptable.
  Patients are followed every 3 months for the first year, every 6 months for the next 4 years, then annually until death.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have recurrent glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of irinotecan in the treatment of patients with recurrent glioma. II. Assess the toxicities of irinotecan in these patients. III. Correlate the pharmacological parameters with toxicity and response to therapy.

OUTLINE: This is a two arm study. Patients are stratified according to prior nitrosourea administration. Patients are assigned to 1 of 2 arms, with only 1 arm being open at any time. Patients assigned to arm I receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22. This is followed by a 2 week rest and continues for a maximum of 6 courses. Patients assigned to arm II receive irinotecan on day 1 every 3 weeks for up to 12 courses. Patients in both arms who received prior nitrosoureas receive reduced starting doses of irinotecan. The dosages may be increased once per patient after the first course if toxic effects are acceptable. Arm I closed as of 10/98, Arm II open as of 10/98. Patients are followed every 3 months for the first year, every 6 months for the next 4 years, then annually until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primary brain glioma Astrocytoma Gliosarcoma Oligodendroglioma Oligoastrocytoma Tumor progression by CT scan or MRI following radiotherapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 3 times upper limit of normal No prior Gilbert's syndrome Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No history of myocardial infarction within 6 months No congestive heart failure requiring therapy Other: No concurrent active second malignancy No uncontrolled infection No other severe concurrent disease Not pregnant or lactating Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior adjuvant chemotherapy regimen and 1 for recurrence (Gliadel is considered 1 regimen) At least 4 weeks since prior chemotherapy At least 6 weeks since prior nitrosoureas No prior irinotecan, topotecan, or aminocamptothecin Endocrine therapy: At least 2 weeks on fixed dose of corticosteroids (or no corticosteroids) prior to baseline scan Radiotherapy: At least 8 weeks since prior radiotherapy Surgery: No surgical resection between last radiotherapy or chemotherapy and study therapy, unless unequivocal tumor growth since surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1998-01; Primary Completion 2001-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan C. Buckner, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Santisteban M, Buckner JC, Reid JM, Wu W, Scheithauer BW, Ames MM, Felten SJ, Nikcevich DA, Wiesenfeld M, Jaeckle KA, Galanis E; North Central Cancer Treatment Group. Phase II trial of two different irinotecan schedules with pharmacokinetic analysis in patients with recurrent glioma: North Central Cancer Treatment Group results. J Neurooncol. 2009 Apr;92(2):165-75. doi: 10.1007/s11060-008-9749-4. Epub 2008 Dec 10. PMID 19066728
- [Result] Laack NN, Ballman KV, Brown PB, O'Neill BP; North Central Cancer Treatment Group. Whole-brain radiotherapy and high-dose methylprednisolone for elderly patients with primary central nervous system lymphoma: Results of North Central Cancer Treatment Group (NCCTG) 96-73-51. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1429-39. doi: 10.1016/j.ijrobp.2006.03.061. PMID 16863926